CLINICAL TRIAL: NCT07383779
Title: Targeted Hypothermia Versus Targeted Normothermia After Convulsive Refractory Status Epilepticus: a Multicenter Randomized Controlled Trial
Brief Title: Targeted Hypothermia Versus Targeted Normothermia After Convulsive Refractory Status Epilepticus
Acronym: HYBERNATUS II
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, LEGRIEL stephane, Investigator Coordinator, Versailles Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P21/14 _ HYBERNATUS_II; 2023-A01518-37 (Other: ID RBC)
Record Dates: First submitted 2025-12-05; First posted 2026-02-03 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Convulsive Refractory Status Epilepticus; Status Epilepticus
MeSH Terms: conditions — Status Epilepticus | interventions — Hypothermia, Induced

STUDY DESIGN:
Intervention Model Description: Intervention group : Targeted temperature management in hypothermia at 33°C [32-34°C] for 24 hours, then progressive rewarming to normothermia 37°C [36.5-37.5°C] up to 72 hours after convulsive refractory SE onset Comparator group : Targeted normothermia 37°C [36.5-37.5°C] for 72 hours after convulsive refractory SE onset
Who Masked: Outcomes Assessor
Masking Description: Discharged patients will receive a centralized phone call interview by an independent assessor blinded of allocation arms at 90 days after randomization to assess GOS-E status (multiple primary outcome). Continuous EEG recordings will be posteriori reviewed by an adjudication committee, composed of three independent neurophysiologist blinded of allocation arms, for identification of patients with progression to electrographic SE (multiple primary outcome).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Targeted Hypothermia (Experimental): Targeted temperature management in hypothermia at 33°C [32-34°C] for 24 hours, then progressive rewarming to normothermia 37°C [36.5-37.5°C] up to 72 hours after convulsive refractory SE onset
  Interventions: Device: Targeted Hypothermia
- Targeted normothermia (No Intervention): Targeted normothermia 37°C [36.5-37.5°C] for 72 hours after convulsive refractory SE onset

INTERVENTIONS:
Device: Targeted Hypothermia — The objective is to lower the core body temperature to 33°C [32-34°C] rapidly after randomization then to maintain this temperature for 24 hours. The management in the targeted hypothermia group will include the following:
  * Sedation with Propofol maintenance infusion at a rate of 2-5 mg/kg/h
  * Hypothermia induction and maintenance using a non-invasive loop-feedback TTM device associating pads directly adhering to the patient's skin (Artic Sun TM provided by the study, similar in all participating centers).
  * Shivering will be assessed using the Bedside Shivering Assessment Scale (BSAS) (Appendix 14) with a tiered approach and avoiding continuous neuromuscular blockade use.
  * After 24 h of targeted hypothermia, rewarming will be standardized at a slow rate of 0.3°C per hour; if used, CisPropofol is progressively decreased (20% every 4 hours) to the lowest dose needed to ensure tolerance of the endotracheal tube
  Arms: Targeted Hypothermia

SUMMARY:
The HYBERNATUS-II study is a phase-III, open-label, randomized controlled trial in patients with convulsive refractory SE receiving mechanical ventilation. Patients are allocated at random to either early targeted hypothermia for 24 hours or targeted normothermia at the acute phase of ICU management. This trial is a superiority multicentric trial and patients will be randomized in a 1:1 ratio using an electronic Cas Report Form.

Before any examination or intervention related to the study may be carried out, the investigator must obtain the freely given, informed and written consent of the participant, or of his/her substitute decision maker (family member, close relative or legal representative) where applicable. However, eligible subjects are unconscious and inherently not able to consent.

Two situations of inclusion are therefore envisaged:

- In case a substitute decision maker is present or contactable: a freely given, informed and written consent of the substitute decision maker will be performed.

- In case a substitute decision maker is not present or contactable in the inclusion time frame, the patient may be included through a process of differed consent. Substitute decision maker will be informed as soon as possible and a freely given, informed and written pursuit consent will be performed.

In all cases, the patient will have to confirm his participation to the study through a freely given, informed and written pursuit consent as soon as their condition allows it. If the patient is under curatorship, the pursuit consent may be given based on his or her own decision. If the patient is under guardianship, the written guardian's consent will also be required.

Individuals liable to participate in studies stipulated in line 1° of article L. 1121-1 of the Code de la Santé Publique (French Public Health Code) benefit from a preliminary medical examination adapted to the study.

Patients will be included after informed consent as soon as possible once they satisfied all eligibility criteria. The inclusion window is until 3.5 hours (210 minutes) after convulsive SE onset. Consecutive eligible patients will be included and randomly allocated in a 1:1 ratio to one of the two procedure groups.

Randomization and concealment will be ensured by using a secure, computer-generated, interactive, response system accessible via the Internet available at each study centre 24H/24. Randomization list will be prepared by an independent statistician who will not be in charge of the analysis. Randomization lists will be generated by a dedicated computer program, with randomly varying sized blocks, and stratified as follows: according to sites, previous history of epilepsy [yes or not], and results of brain imaging [Abnormal Brain Imaging or not].

Each investigator will be able to access the randomization site using a personal password.

Randomization will be carried out after checking of the inclusion criteria and the absence of exclusion criteria and after obtaining a written and informed consent or according to the emergency procedure by the principal investigator or a physician representing the investigator before the person is enrolled in the study of each centre involved in the study. Each patient will be assigned a unique identification number. An inclusion confirmation will be sent by email to the investigator specifying the allocated procedure arm.

Patients will be randomly allocated to one of the two study procedure groups.

The two groups will differ only in the administration of early targeted hypothermia for 24 hours or targeted normothermia at the acute phase of ICU management. All other treatment will be standardized in the two groups.

Targeted Hypothermia group : Implementation of allocation arm is started within 30 min after randomization.The objective is to lower the core body temperature to 33°C [32-34°C] rapidly after randomization then to maintain this temperature for 24 hours. The management in the targeted hypothermia group will include the following.

Targeted normothermia group. Implementation of allocation arm is started within 30 min after randomization. The objective of the control group is to ensure normothermia 37° [36.5-37.5°C] for 72 hours after randomization. Antipyretic treatments will be given in case of a core temperature higher than 37.8°C. In case of failure, cooling with a surface non-invasive loop-feedback TTM device associating pads directly adhering to the patient's skin (Artic Sun TM provided by the study, similar in all participating centers) will be initiated with a target temperature of 37° [36.5-37.5°C]. No active warming will be provided for patients in the normothermia group who had a spontaneous body temperature below 36.5°C.

Patients included in the study will be followed until the 90th day after inclusion. The duration of the participation will therefore be 3 months for each patient.

DETAILED DESCRIPTION:
The HYBERNATUS-II trial is a continuation of the collaboration of the previously published HYBERNATUS trial1 supplemented by new collaborations from the ICTALGROUP research network (https://ictalgroup.org).

The HYBERNATUS trial (NCT01359332) was a multicenter, open-label, outcome assessor-blinded, parallel-group, randomized, controlled trial in patients with convulsive status epilepticus (SE) requiring admission to the intensive care unit (ICU) and mechanical ventilation. The main goal of the HYBERNATUS trial was to determine whether therapeutic hypothermia 33°C [32-34°C] for 24 hours has neuroprotective effects compared to standard care alone. The trial showed no significant benefit with respect to good functional outcome from the addition of therapeutic hypothermia to standard antiseizure therapy: a maximum Glasgow Outcome Scale (GOS) score of 5 occurred in 67 of 138 patients (49%) in the hypothermia group and in 56 of 130 patients (43%) in the control group (odds ratio, 1.22; 95% confidence interval (CI), 0.75 to 1.99; P=0.43).

The HYBERNATUS-II study is a phase-III, open-label, randomized controlled trial in which a targeted hypothermia [targeted temperature management (TTM) at 33°C [32-34°C] in patients with convulsive refractory SE will be compared with targeted normothermia 37°C [36.5-37.5°C] (See more details of objectives in Sections 4.1 and 4.2). Patients eligible for inclusion will be unconscious adult patients aged from 18 to 65 years with convulsive refractory SE receiving mechanical ventilation (See more details for inclusion in Sections 5.1 and 5.2).

Consent will be obtained from a substitute decision maker as eligible subjects are unconscious and inherently not able to consent. Thus, the patient will have to confirm his participation to the study as soon as their condition allows for informed consent. Patients who are eligible but incapable of receiving information and for whom substitute decision maker is not present or contactable may be included through a process of differed consent. Substitute decision maker will be informed as soon as possible, and patient will be informed about participation as soon as their clinical status allows. In this case, substitute decision maker's and/or patient's written consent will be obtained as soon as possible. (See more details for ethical considerations in Sections 11.0). Once consent obtained, patients will be included and randomized in one of the two following allocation arms: targeted hypothermia at 33°C [32-34°C] or targeted normothermia 37°C [36.5-37.5°C]. Randomization will be centralized and stratified according to sites, previous history of epilepsy [yes or not], and results of brain imaging [Abnormal Brain Imaging or not]. The two groups will differ only in the administration of TTM at 33°C [32-34°C] or normothermia during the first 24 hours. For the targeted hypothermia group: the temperature will be rapidly decreased and maintained at 33°C [32-34°C] for 24 hours using servo-regulated temperature management devices. Thus, patients will be progressively rewarmed and maintained at normothermia for a total of 72 hours of temperature targeted management. For the normothermia group: patients will be maintained at normothermia 37°C [36.5-37.5°C] for 72 hours.

The choice of TTM at 33°C has been guided by the experimental data indicating dual neuroprotective and antiseizure effects of hypothermia, and the compromise of tolerance of moderate hypothermia in humans.2,3 The duration of 24 hours for targeted hypothermia can be argued by the experience of safety and preliminary data coming from the HYBERNATUS trial1, and the recommended timeframe of seizure suppression (cessation of electrographic seizures or suppression burst).4,5 In both treatment groups, anesthetic agent will be Propofol, a powerful antiseizure agent with a short half-life, at a maximal rate of 5 mg/kg/hour for the maximal duration of 48 hours, minimizing the time of sedation and the risk of Propofol related infusion syndrome. All other treatments will be standardized in the two groups. Anesthetic withdrawal will be progressively performed according to the half-life of Propofol to avoid the risk of Super Refractory Status Epilepticus.

Patients will be continuously monitored for core temperature (bladder or esophageal probes) and continuous electroencephalography (cEEG) during the first 72 hours of management in both groups. In both allocation arms, the therapeutic goal will be seizure suppression. Patients will be followed-up daily from randomization to day 3, then periodically at day-7, day-14, day-28, ICU/hospital discharge and day-90. In addition to the usual demographic data, the data collected will relate to comorbidities, the current clinical history, cause of convulsive refractory SE, treatments and anesthetics received, core temperature every hour during the first 72 hours, performed diagnostic procedures, the observed adverse events and the various parameters allowing the calculation of different severity and organ failure scores (Simplified Acute Physiology Score 2 (SAPS 2), Logistic Organ Dysfunction score (LODs)) at baseline and up to ICU discharge.

Patients receiving targeted hypothermia will be closely monitored for adverse effects such as infections, and Propofol related infusion syndrome will be carefully checked in both allocation arms.

Discharged patients will receive a centralized phone call interview by an independent assessor blinded of allocation arms at 90 days after randomization to assess GOS-E status (multiple primary outcome). Continuous EEG recordings will be posteriori reviewed by an adjudication committee, composed of three independent neurophysiologist blinded of allocation arms, for identification of patients with progression to electrographic SE (multiple-primary outcome). Follow-up will be censored at day-90.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years [18-65 years]
* Continued motor seizure activity lasting more than 5 minutes, or two or more motor seizures without a return to baseline level of consciousness in the interval at least 5 minutes after the first seizure
* Refractory to two recommended antiseizure medications (benzodiazepine and "classic" antiseizure drug)
* Receiving mechanical ventilation
* Time from seizure onset no longer than 3.5 hours (210 min)
* Consent to participate (patient's relative or emergent consent)

Exclusion Criteria:

* Estimated pre-morbid GOS-E score < 5
* Preexisting ultimately fatal comorbidity < 1 year
* Patients unlikely to survive for the next 24 hours
* Full recovery at time of inclusion
* Need for emergent surgery or interventional neuroradiology for bleeding embolization (neurosurgery or other precluding therapeutic hypothermia)
* Postanoxic status epilepticus
* Traumatic Brain Injury with an acute bleeding on Computed Tomographic (CT) scan or Magnetic Resonance Imaging (MRI) of the brain
* Bacterial meningitis as a cause of convulsive SE
* Cryoglobulinemia, sickle cell disease, serum cold agglutinins comorbidities
* Pregnancy
* Absence of coverage by the French/European statutory healthcare insurance system

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 466 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of TH 33°C [32-34°C] for 24 hours in improving the 90-day neurological outcome | 90 days
  Percentage of patients who reached the level [5-8] of the GOS-E scale [scale range 1-8, 8 best score] in each group at day 90
Decreasing post-randomization progression to electrographic SE at day-1 in patients with RSE | 1 day
  Percentage of patients experiencing progression to electrographic SE (from 1 to 25 hours after randomization)

SECONDARY OUTCOMES:
To assess the efficacy of TH on reducing the burden of drugs | 1 day
  Total weight-based dose of propofol and other anesthetic agent(s) simultaneously used between 1 to 25 hours after randomization (mg/kg each)
To assess the efficacy of TH on reducing the burden of seizures on day 1 | 1 day
  Electroencephalographic seizure (ictal) burden in minutes at day 1 (1 to 25 hours after randomization)
To assess the efficacy of TH reducing the burden of seizures on day 2 and 3 | 2 and 3 days
  Percentage of patients with super refractory SE at day 2 and/or 3 after randomization: 1) ongoing seizures despite 24 hours or more after onset of anesthetic therapy (e.g., Propofol), or 2) recurrence of seizures upon reduction or withdrawal of therapeutic anesthetic coma
To assess the tolerance of the intervention (pneumonia) | 7 days
  Percentage of patients with pneumonia requiring antibiotherapy between day-1 and day-7 after randomization
To assess the tolerance of the intervention (other infections) | 7 days
  Percentage of patients with infection requiring the use of antimicrobial agent between day-3 and -7 after randomization
To improve the short, mid-term outcomes (inotropic and/or vasopressor) | day-1, -2 and -3 after randomization
  Percentage of patients with inotropic and/or vasopressor at day-1, -2 and -3 after randomization
To improve the short, mid-term outcomes (mechanical ventilation) | day-1, -2 and -3 after randomization
  Mechanical ventilation duration defined by time (in days) between extubation and intubation times (after randomization)
To improve the short, mid-term outcomes (Coma-free days ) | day-1, -2 and -3 after randomization
  Coma-free days during hospitalization defined by total hospital length of stay without coma after randomization (in days)
To improve the short, mid-term outcomes (ICU mortality) | 90 Days
  Percentage of deaths at ICU discharge
To improve the short, mid-term outcomes (hospital mortality) | 90 Days
  Percentage of deaths at hospital discharge
To improve the short, mid-term outcomes (90-day mortality) | 90 Days
  Percentage of deaths at day-90 after randomization
To improve the short, mid-term outcomes (Physical/functional) | 90 Days
  Barthel index and FSS scores at day 90 after randomization
To improve the short, mid-term outcomes (cognitive ) | 90 Days
  TICS-m score at day 90 after randomization
To improve the short, mid-term outcomes (mental health status) | 90 Days
  HADS and IES-R scores at day 90 after randomization
To improve the short, mid-term outcomes (return to work) | 90 Days
  WPAI-GH score at day 90 after randomization
To improve the short, mid-term outcomes (Quality-of-life) | 90 Days
  SF36 score at day 90 after randomization

CONTACTS AND LOCATIONS:
Locations (20):
- France (20):
  - Hôpital Ambroise Paré, Boulogne-Billancourt
  - CHU Brest, Brest
  - CH Simone Veil, Cannes
  - Hôpital Louis Mourier, Colombes
  - CH Sud Francilien, Corbeil-Essonnes
  - CHU Dijon, Dijon
  - CH Versailles, Le Chesnay
  - CH Le Mans, Le Mans
  - Hôpital de la Croix-Rousse, Lyon
  - Hôpital Edouard Herriot, Lyon
  - CH Melun-Sénart, Melun
  - CH Annecy Genevois, Metz-Tessy
  - CHU Nantes, Nantes
  - CHR Orléans, Orléans
  - GH Paris Saint-Joseph, Paris
  - Hôpital COCHIN, Paris
  - CHU Rennes, Rennes
  - Hôpital Hautepierre, Strasbourg
  - Hôpital Foch, Suresnes
  - CHITS Toulon, Toulon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Legriel S. Hypothermia as a treatment in status epilepticus: A narrative review. Epilepsy Behav. 2019 Dec;101(Pt B):106298. doi: 10.1016/j.yebeh.2019.04.051. Epub 2019 May 24. PMID 31133509
- [Background] Legriel S. Hypothermia as an adjuvant treatment in paediatric refractory or super-refractory status epilepticus. Dev Med Child Neurol. 2020 Sep;62(9):1017-1023. doi: 10.1111/dmcn.14562. Epub 2020 May 15. PMID 32412660
- [Background] Legriel S, Fontaine C, Jacq G. The value of hypothermia as a neuroprotective and antiepileptic strategy in patients with status epilepticus: an update of the literature. Expert Rev Neurother. 2025 Jan;25(1):57-66. doi: 10.1080/14737175.2024.2432869. Epub 2024 Nov 24. PMID 39582132
- [Background] Legriel S, Lemiale V, Schenck M, Chelly J, Laurent V, Daviaud F, Srairi M, Hamdi A, Geri G, Rossignol T, Hilly-Ginoux J, Boisrame-Helms J, Louart B, Malissin I, Mongardon N, Planquette B, Thirion M, Merceron S, Canet E, Pico F, Tran-Dinh YR, Bedos JP, Azoulay E, Resche-Rigon M, Cariou A; HYBERNATUS Study Group. Hypothermia for Neuroprotection in Convulsive Status Epilepticus. N Engl J Med. 2016 Dec 22;375(25):2457-2467. doi: 10.1056/NEJMoa1608193. PMID 28002714